CLINICAL TRIAL: NCT06877767
Title: Effects of Graston Versus Active Release Technique on Hamstring Flexibility, Pain and Disability in Females With Non Specific Low Back Pain
Brief Title: Graston Versus Active Release Technique in Females With Non Specific Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0148
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
Keywords: disability evaluation; females; low back pain; pain assessment; Range of motion; Soft tissue
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: graston technique (Experimental): Group A: baseline physical therapy treatment along with graston technique
  Interventions: Other: Graston Technique
- Group B: active release technique (Active Comparator): Group B: baseline physical therapy treatment along with active release technique
  Interventions: Other: Active Release Technique

INTERVENTIONS:
Other: Graston Technique — Following the conventional treatment, this technique will be carried out through Graston tool called "GT-1" The special Graston Emollient or lubricant will be applied to the hamstrings of the subject then the tool used to find adhesions and break them up for 2.5 minutes per leg. First, the subject will lay prone and bent the knee joint to around 30° to 60°.The Graston instrument will be rubbed on each subject 30 times for 60 seconds from the gluteal line to the popliteal fossa. This treatment technique will be applied twice a week
  Arms: Group A: graston technique
Other: Active Release Technique — Following the conventional treatment, subject received single session of ART on each side. There are 3 steps to perform ART. Step 1:Subject lies supine on the plinth and gentle tension was applied to the hamstring muscle along the entire length while stretching the leg in different positions to better work the muscle. Step 2: Gentle tension will be applied at the origin and insertion of the hamstring muscle. Step 3: The therapist will place tension on the bellies of hamstrings longitudinally at a specific tension & ask the patient to extend his knee as per ART protocol.• This is done for 2.5 minutes on each leg. • This treatment technique will be applied twice a week.
  Arms: Group B: active release technique

SUMMARY:
Non-specific Low Back Pain defined by tension, soreness, and/or stiffness of the lower back with unknown origins of pain. Reduction in hamstrings flexibility has found to be one of the causes for development of low back pain. Soft tissue manipulation can help loosen these muscles up and decrease a lot of the pain an individual may be having. Two specific kinds of soft tissue techniques will be utilized in this study are Graston Technique and Active Release Technique. So the aim of this project is to compare the effects of Graston Technique (GT) and Active Release Technique (ART) in the females with NSLBP. The study will be a randomized clinical trial and will be conducted in Allama Iqbal Memorial Teaching Hospital Sialkot. Non-probability convenience sampling technique will be used and participants will be recruited in groups after randomization. The subjects (n=40) will be divided into two groups. First group will include 20 women and graston technique will be applied. Group B will include 20 women and receive active release technique. Both the Groups will receive Hot Pack for 10 minutes, Passive stretching and Therapeutic Exercises for core stability; will be performed 2 times a week with 10 second hold of each exercise. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Universal Goniometer (GU) for Active knee extension test and popliteal angle measurement and Oswestry Disability Index for disability in the female patients with NSLBP. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

DETAILED DESCRIPTION:
Low back pain (LBP) is a condition experienced at least once by more than 80% of the human race the world over. More than 85% of cases of LBP in the USA are classified as nonspecific LBP defined by tension, soreness, and/or stiffness of the lower back with unknown origins of pain. Non-specific low back pain (NLBP) or "simple backache" is characterized as an LBP not due to any identifiable disease such as nerve root pain and severe spinal pathologies such as infection, tumor, osteoporosis, rheumatoid arthritis, fracture or inflammation. Back pain causes decreased lumbar extensibility, limited range of motion (LOM) and gait ability, and change of rhythm in the pelvis, limitations that can restrict social activities. One of the most widely studied outcomes in LBP patients is the reduction of hamstring extensibility. A shortening of the hamstring may result in LOM of the knee joint, restricting a person's ability to walk and run. In addition, it increases posterior pelvic tilting and reduces lumbar lordosis, contributing to a flat back that can result in low back. Methods for increasing the length of the shortened hamstring include stretching, eccentric resistance exercise, Graston instrument soft tissue mobilization, and self-myofascial release. Hamstring tightness is prevalent with the low back pain yet there is a need to establish a standardized treatment protocol for the condition. That's why this study will try to find out effective manner to release the pain and improve the flexibility of hamstring muscles.

The aim of this study is to determine the comparative effects of ART and Graston Technique specifically with each other on Hamstring flexibility, pain and disability in females with nonspecific low back pain. Therefore, this study will put into effect so that Graston Technique and ART can be compared against each other to see if one is more effective for restoration of full soft tissue function and relieving pain. This study will provide significant information that will aid in the creation of therapeutic interventions to improve pain, range of motion and functional limitations in females with non-specific low back pain. Graston Technique (GT) is a soft tissue mobilization treatment method using a tool that generates mechanical micro-traumatic damage to the treated area. In ART the goal is to remove the soft tissue adhesions by decreasing tissue tension. The muscle is taken from a shortened position to a lengthened position while a contact hand is holding tissue tension longitudinally along the soft tissue fibers.

ELIGIBILITY:
Inclusion Criteria:

* Females with Non Specific Low Back Pain
* Age group between 25 and 50 years
* History of NSLBP for at least 3 months
* Popliteal angle Numeric Rating Scale (NRS) score of 3-7/10
* The Oswestry Disability Index (ODI) score of 20-60
* Patients agree to sign written consent form.

Exclusion Criteria:

* Acute onset of pain and pain with radiation below knee.
* Any history of injury in the lower extremity in the past three months.
* Constant or persistent severe pain, inflammatory conditions (rheumatoid arthritis, ankylosing spondylitis)
* participants must not be taking any treatment of a musculoskeletal nature.
* Any previous surgery around the knee and hip
* hamstrings injury and strains
* Pregnant females
* Allergy to hot pack

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  The NPRS is a standardized self-report device consisting of a horizontal line used to estimate the subjective level of pain intensity. It is a 10 Points numerical scale, corresponding to the degree of pain. 1 being least level of pain and 10 being the highest level of pain.
Oswestry Disability Index | 4 weeks
  Oswestry Disability Questionnaire will be used for measuring the level of disability in patients with low back pain. This questionnaire consists of 10 categories, each of which score on scale of 0-5, where 0 shows no disability and 5 shows the greatest disability. Each section caries 05 Questions describing minimum to maximum level of disability. The test is considered the 'gold standard' of low back functional outcome tools. It has 10 different sections. For each section the total possible score is 5. If all 10 sections are completed the score is calculated and interpreted in percentage measures.
Universal Goniometer (UG) | 4 weeks
  Universal Goniometer (UG) is used for the measurement of popliteal angle and active knee extension test. To measure the popliteal angle, an active knee extension test will be applied. The the testing limb in 90º hip and knee flexion and the non testing limb in an extended with the subject supine on plinth, with the help of goniometer angle is measured between thigh and calf. For AKE test participants are positioned supine on a plinth. From this position, subjects are instructed to extend the knee until they felt a strong resistance, holding this final position for 2 to 3 seconds to allow the goniometric reading .

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Allama Iqbal Memorial Teaching Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allam NM, Eladl HM, Elruwaili LT, Elruwaili LF, Elbenya TJ, Elanzi EM, Elquobisi FF, Elgadoa HM, Elghaleb MA, Elsaeid MS, Elquarenes RA, Elrashed SM, Elmobarak SS, Elkholi SM, Eid MM, Alanazi AM, Nambi G, Abdelbasset WK. Correlation between hamstring muscle tightness and incidence of low back pain in female students at Jouf University, Saudi Arabia. Eur Rev Med Pharmacol Sci. 2022 Nov;26(21):7779-7787. doi: 10.26355/eurrev_202211_30127. PMID 36394725
- [Background] Sassonker K, Magnezi R, Moran D. Comparing right and left hamstring flexibility and its association to nonspecific lowr back pain among women of different age groups. J Bodyw Mov Ther. 2023 Oct;36:404-409. doi: 10.1016/j.jbmt.2023.07.014. Epub 2023 Sep 9. PMID 37949592
- [Background] Hori M, Hasegawa H, Takasaki H. Comparisons of hamstring flexibility between individuals with and without low back pain: systematic review with meta-analysis. Physiother Theory Pract. 2021 May;37(5):559-582. doi: 10.1080/09593985.2019.1639868. Epub 2019 Jul 18. PMID 31317831
- [Background] Nazary-Moghadam S, Yahya-Zadeh A, Zare MA, Ali Mohammadi M, Marouzi P, Zeinalzadeh A. Comparison of utilizing modified hold-relax, muscle energy technique, and instrument-assisted soft tissue mobilization on hamstring muscle length in healthy athletes: Randomized controlled trial. J Bodyw Mov Ther. 2023 Jul;35:151-157. doi: 10.1016/j.jbmt.2023.04.079. Epub 2023 Apr 21. PMID 37330762
- [Background] Moon JH, Jung JH, Won YS, Cho HY. Immediate effects of Graston Technique on hamstring muscle extensibility and pain intensity in patients with nonspecific low back pain. J Phys Ther Sci. 2017 Feb;29(2):224-227. doi: 10.1589/jpts.29.224. Epub 2017 Feb 24. PMID 28265144